CLINICAL TRIAL: NCT07112391
Title: Invasive Hemodynamic Study of Structural Heart Diseases: A Monocentric, Non-Randomized Approach
Brief Title: Pressure-Volume Loop Assessment in Valvular Heart Disease
Acronym: VHD-PV-loop
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0116
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Structural Heart Disease; Interventional Cardiology
Keywords: Chronic heart failure; Structural heart disease; Interventional cardiology; Multimodality imaging
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe valvular heart disease: Patients with severe Valvular Heart Disease (VHD) will undergo a RV volumetric assessment (MRI, CT, 3D-echocardiography) followed within 72h by an invasive assessment of RV-PA coupling using conductance catheters, either as a preoperative evaluation or at the time of transcatheter valvular intervention. Echocardiographic images will be acquired during right heart catheterization (RHC) in order to be compared to the gold-standard.
  Interventions: Other: Observational Invasive Hemodynamic Assessment

INTERVENTIONS:
Other: Observational Invasive Hemodynamic Assessment — Collection and analysis of invasive hemodynamic data obtained through routine cardiac catheterization performed as part of standard care. No intervention is mandated by the study protocol.
  Other Names: Cardiac Catheterization; Hemodynamic Procedure

SUMMARY:
The VHD PV loop study intends to assess invasive right ventricular to pulmonary artery (RV-PA) coupling in patients with valvular heart disease (VHD). Invasive RV-PA coupling is measured by using conductance catheters, the gold standard assessment for ventricular physiology. Several non-invasive parameters have been reported as surrogates for this complex physiological entity, but none of them has been tested against the gold-standard in this population. Based on this, our main objective is to assess the correlation of imaging derived RV-PA coupling in comparison to the invasive measurement.

DETAILED DESCRIPTION:
This study aims to improve the assessment of right ventricular (RV) function in patients with valvular heart disease (VHD), by validating non-invasive imaging parameters of right ventricular to pulmonary artery (RV-PA) coupling against invasive measurements using conductance catheters-the gold standard for evaluating RV hemodynamics.

Currently available non-invasive tools do not always provide reliable evaluation of RV-PA coupling. This study seeks to identify accurate imaging surrogates to support clinical decision-making, particularly in conditions such as secondary mitral regurgitation, tricuspid regurgitation, and right-sided structural heart disease.

By correlating non-invasive indices-such as tricuspid annular plane systolic excursion to pulmonary artery systolic pressure ratio (TAPSE/PASP) and RV strain-with invasive data, the study may enhance diagnostic strategies, improve patient care, and support future prognostic and therapeutic investigations. Data may also contribute to post hoc analyses in existing registries and help refine our understanding of RV adaptation in structural heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old);
* Patients with severe structural heart disease (meeting at least one of the following three criteria):

  * Heart failure with moderate-to-severe or severe secondary mitral regurgitation
  * At least severe tricuspid regurgitation
  * Significant pulmonary valve stenosis and/or regurgitation

Exclusion Criteria:

* Patients under legal guardianship or protection (e.g., guardianship, trusteeship, or any other legal protection measure);
* Pregnant or breastfeeding women;
* Vulnerable individuals (e.g., persons deprived of liberty, adults under legal protection);
* Contraindication to right heart catheterization, including:

  * Known proximal venous occlusion of the superior or inferior vena cava territory
  * Presence of a mobile mass in the right heart chambers
  * Significant tricuspid stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients referred to Nantes University Hospital for the treatment of significant VHD.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2027-09-04 (Estimated)

PRIMARY OUTCOMES:
Correlation with non-invasive echocardiographic parameters | During right heart catheterization (Day 1)
  Assessment of diagnostic performances of TAPSE/PAPS, RVFWLS/PAPS and FAC/PAPS ratios compared to Ees/Ea ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Robin LE RUZ, MD, PhD, Principal Investigator — Hospital of Nantes
Locations (1):
- CHU of NANTES, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided